CLINICAL TRIAL: NCT01250444
Title: Inspiratory Muscle Training: Effects on Blood Pressure, Heart Rate Variability and Functional Capacity in Hypertensive Patients.
Brief Title: Effects of Inspiratory Muscle Training on Cardiovascular Function in Hypertension.
Acronym: TREMVEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Pedro Dal Lago, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TREMVEN
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-10

CONDITIONS: Reduction of Blood Pressure in Hypertensive Patients.; Improvement of Cardiovascular Autonomic Control.; Improvement of Functional Capacity.; Improvement of Quality of Life.
Keywords: Inspiratory Muscle Training; Hypertension; Breathing Exercises; Cardiac Rehabilitation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inspiratory Muscle Training (Experimental): It will me performed a loaded training of ventilatory muscles in patients with Hypertension. Its is done with the practice of breathing exercises associated to an training device, specific for this kind of intervention.
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Breathing exercises associated to the use of a training device with predetermined pressure load, daily, 30 minutes per day, during eight weeks.

SUMMARY:
The purpose of this study is to determine inspiratory muscle training effects on blood pressure, functional capacity and quality of life in hypertensive patients.

DETAILED DESCRIPTION:
The interaction between respiratory function and cardiovascular system, as well as the present alterations in these systems, due to diseases such as Hypertension, diabetes and chronic heart failure, are the factors that potentially participate of the pathogenic frame in these situations. Consequently, it is so related to reduction of functional capacity, endothelial dysfunction of the sympathetic and parasympathetic cardiovascular control and morphologic alterations on the skeletal muscles, including ventilatory muscles.

On the other hand, a proinflammatory state also participates of this dysfunction and reduced function capacity situation. Cardiovascular risk factors, such as hypertension, increased heart rate variability, diabetes and heart failure explain the occurrence of the majority of cardiovascular events in the entire world and so in Brazil. Studies with experimental models and in patients with cardiovascular diseases identified important inflammatory activity associated to risk factors and preceding clinical events.

Inspiratory muscle training (IMT) shows consistent results in the improvement of functional capacity in athletes, sedentary subjects, heart failure patients and in animals submitted to an IMT model.

The study of alterations in cardiorespiratory interaction, functional capacity and cardiovascular control mechanisms (sympathetic, parasympathetic by heart rate variability), altogether, in hypertension, is a single opportunity to identify new pathogenic mechanisms involved in the reduction of functional capacity as well as promote its quantification. Therefore, the effects of IMT on these alterations are still not well understood. In this way, the response to IMT is a complement to epidemiologic and clinical models, as potential source of new possibilities in the research field.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 70
2. Hypertension in all stages:

2.1. Prehypertension - Systolic blood pressure (SBP) of 120 to 139 and/or diastolic blood pressure (DBP) of 80 to 89 mmHg 2.2.Stage 1 Hypertension - SBP of 140 to 159 mmHg and/or DBP of 90 to 99 mmHg 2.3.Stage 2 Hypertension - SBP ≥ 160 mmHg and/or DBP ≥ 100 mmHg

Exclusion Criteria:

1. Disagreement with consent form
2. Thoracic pain (angina)
3. Hypertension instability
4. Antihypertensive drugs alterations within 30 days before or during the study
5. Diabetes
6. Chronic pulmonary obstructive disease
7. Incapability of executing the functional tests
8. Asthma
9. Chronic Heart Failure
10. Obesity
11. Cardiovascular diseases complications

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Differences on blood pressure levels | eight weeks
  Blood pressure behavior is accessed by Ambulatory Blood Pressure Monitorying.

SECONDARY OUTCOMES:
improvement of Heart rate variability | eight weeks
improvement of quality of life | eigth weeks
  To measure the quality of life, it is used the SF36 short form questionary.
Improvement of Functional Capacity | eight weeks
  It is measure by the oxytgen consumption accessed by ergospirometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro Dal Lago, Porto Alegre, Rio Grande do Sul, Brazil